CLINICAL TRIAL: NCT00456729
Title: Malabsorption as a Cause of Iron Treatment Failure in Infants - A Clinical Observational Study
Brief Title: Malabsorption as a Cause of Iron Treatment Failure in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4150905.EMC
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-01

CONDITIONS: Iron Deficiency; Malabsorption
Keywords: Iron deficiency; Malabsorption; Giardiasis
MeSH Terms: conditions — Iron Deficiencies; Malabsorption Syndromes; Giardiasis | interventions — Metronidazole; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Metronidazole
Procedure: Blood tests

SUMMARY:
Infants should receive prophylacatic iron supplementation since age 4 months till one year. Patients suffering from malabsorption, mainly Giardia infestation may develop iron deficiency resistent to further iron treatment. The purpose of this study is to assess the incidence of malabsorption in those infants and to examine the results of empiric treatment with metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* All infants referred to the Pediatric Hematology Unit because lack of response to iron treatment.

Exclusion Criteria:

* Patients diagnosed with specific malabsorption causes like Celiac or Cystic Fibrosis.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2006-05; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hgb level

SECONDARY OUTCOMES:
Iron level
Ferritin Level

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center; Tania Hanchis, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel